CLINICAL TRIAL: NCT00694525
Title: Potential Modulatory Role of Osteoprotegerin in Bone Metabolism of Patients With 21-Hydroxylase Deficiency
Brief Title: Role of the Protein Osteoprotegerin in the Bone Health of Women With Congenital Adrenal Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Office of Rare Diseases (ORD) (NIH)
Responsible Party: Maria I. New, MD, Mount Sinai School of Medicine
Other Study IDs: RDCRN 5611
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: 21OHD; 21-hydroxylase deficiency; CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — With participant's permission, 5 mL of blood will be stored for potential new blood markers in the future.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women in this group will have 21-OHD CAH.
- 2: Women in this group will be healthy controls and will not have 21-OHD CAH.

SUMMARY:
21-hydroxylase deficiency (21-OHD) is an inherited disorder that results from a mutation on the CYP21A2 gene. It affects the adrenal glands and is the most common cause of congenital adrenal hyperplasia (CAH). 21-OHD CAH causes the body to produce an insufficient amount of cortisol and an excess of androgen, the type of hormone that produces male characteristics. The primary treatment for 21-OHD CAH, glucocorticoid replacement therapy, has been shown to cause bone loss. However, the elevated hormone levels caused by 21-OHD CAH may increase production of the protein osteoprotegerin (OPG), which in turn may protect against bone loss. This study will compare bone density and OPG levels in women who have 21-OHD CAH and have undergone a lifetime of glucocorticoid replacement therapy to that in women who have neither of these criteria. In doing so, the study will aim to determine the relationship between OPG and bone loss.

DETAILED DESCRIPTION:
Because of the excess of androgen caused by 21-OHD CAH, women with CAH may exhibit some male-like characteristics. Glucocorticoids are a member of a class of drugs called corticosteroids, which are used in hormone replacement therapy. In order to counteract the effects of 21-OHD CAH, women with the disease are given hormone replacement therapy with glucocorticoids beginning at infancy. Glucocorticoids are known to cause bone loss. Despite many years of treatment with glucocorticoids, however, young women with 21-OHD CAH seem to be protected against bone loss. Researchers believe that the increased androgen levels in these women leads to increased estrogen levels, which in turn increases OPG production. The increase in OPG levels may protect women against bone loss. This study will evaluate bone density and OPG levels in women with and without 21-OHD CAH to determine the relationship between OPG and bone loss.

Participants in this observational study will attend only one study visit. At this visit, they will undergo a blood draw; a scan of their lower spine, hip, and forearm; height and weight measurements; and a body fat analysis test. This last test will entail a weak and painless electrical signal being sent from foot to foot. Participants will not attend any follow-up visits for this study.

ELIGIBILITY:
Inclusion Criteria:

For People with 21-OHD CAH:

* 21-OHD CAH has been documented by molecular genetic analysis (mutations on CYP21A2 gene on both parental alleles)
* Treatment with glucocorticoid replacement since infancy (begun within the first year)
* Available hormonal data and treatment details over the 5 years prior to study entry
* Premenopausal

For Healthy Controls:

* No diagnosis of 21-OHD CAH, as confirmed by molecular genetic analysis
* No first degree relative is enrolled as a 21-OHD CAHparticipant
* Premenopausal

Exclusion Criteria:

* Medical disorder or treatment with medications known to affect bone density (other than glucocorticoids for 21-OHD CAH patients), including, but not limited to growth hormone, IGF-I, depo-medroxyprogesterone acetate, biphosphonates, oral contraceptives, androgens, thyroxine, or aromatase inhibitors
* Pregnant
* Any smoking within the 6 months prior to study entry
* Cardiac pacemaker or other implanted electronic medical device

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal women between the ages of 20 and 35 who have 21-OHD CAH or do not have 21-OHD CAH.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of levels of OPG | Measured throughout the study

SECONDARY OUTCOMES:
Comparison of bone mineral density | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lin Su, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Canalis E, Bilezikian JP, Angeli A, Giustina A. Perspectives on glucocorticoid-induced osteoporosis. Bone. 2004 Apr;34(4):593-8. doi: 10.1016/j.bone.2003.11.026. No abstract available. PMID 15050888
- [Background] Paganini C, Radetti G, Livieri C, Braga V, Migliavacca D, Adami S. Height, bone mineral density and bone markers in congenital adrenal hyperplasia. Horm Res. 2000;54(4):164-8. doi: 10.1159/000053253. PMID 11416232
- [Background] King JA, Wisniewski AB, Bankowski BJ, Carson KA, Zacur HA, Migeon CJ. Long-term corticosteroid replacement and bone mineral density in adult women with classical congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2006 Mar;91(3):865-9. doi: 10.1210/jc.2005-0745. Epub 2005 Nov 8. PMID 16278269
- [Background] Kudlacek S, Schneider B, Woloszczuk W, Pietschmann P, Willvonseder R; Austrian Study Group on Normative Values of Bone Metabolism. Serum levels of osteoprotegerin increase with age in a healthy adult population. Bone. 2003 Jun;32(6):681-6. doi: 10.1016/s8756-3282(03)00090-5. PMID 12810175
- [Background] Hagenfeldt K, Martin Ritzen E, Ringertz H, Helleday J, Carlstrom K. Bone mass and body composition of adult women with congenital virilizing 21-hydroxylase deficiency after glucocorticoid treatment since infancy. Eur J Endocrinol. 2000 Nov;143(5):667-71. doi: 10.1530/eje.0.1430667. PMID 11078991